CLINICAL TRIAL: NCT03037580
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of Oral Treprostinil in Subjects With Pulmonary Hypertension (PH) in Heart Failure With Preserved Ejection Fraction (HFpEF)
Brief Title: Oral Treprostinil in Subjects With Pulmonary Hypertension Associated With Heart Failure With Preserved Ejection Fraction
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Terminated by sponsor
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDE-HF-301
Record Dates: First submitted 2017-01-27; First posted 2017-01-31 (Estimated); Results first posted 2020-10-22 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Pulmonary Hypertension; Heart Failure With Preserved Ejection Fraction
Keywords: Pulmonary Hypertension; 6-Minute Walk Test; HFpEF; Oral Treprostinil
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — treprostinil; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Oral treprostinil (Experimental): Sustained-release oral tablets for TID administration
  Interventions: Drug: Oral treprostinil
- Placebo (Placebo Comparator): Placebo (sugar pill) for TID oral administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral treprostinil — Sustained-release oral tablets for TID administration
  Other Names: Treprostinil diethanolamine, treprostinil diolamine
  Arms: Oral treprostinil
Drug: Placebo — Placebo (sugar pill) for TID oral administration
  Other Names: Matching placebo (sugar pill)
  Arms: Placebo

SUMMARY:
This was a multicenter, randomized (1:1; oral treprostinil to placebo), double-blind, placebo-controlled study in subjects with World Health Organization (WHO) Group 2 pulmonary hypertension (PH) associated with heart failure with preserved ejection fraction (HFpEF). Once randomized, subjects took the initial dose of study drug at the study site on the day of randomization. Subjects returned to the study site for visits scheduled at Weeks 6, 12, 18, and 24. The duration of study participation was approximately 28 weeks from Screening until study completion (includes a 30-day Screening Phase and 24-week Treatment Phase).

The study was discontinued by the Sponsor on 14 October 2019 due to slow enrollment. As only a small portion of the anticipated total subjects had been enrolled, with many terminating early due to the study termination, there was a limited ability to explore the effect of oral treprostinil in this indication in this study.

DETAILED DESCRIPTION:
Study TDE-HF-301 was a multicenter, randomized, double-blind, placebo-controlled study designed to investigate the effect of oral treprostinil compared with placebo on exercise capacity in subjects with WHO Group 2 PH associated with HFpEF.

Once randomized, subjects were dispensed study drug and took an initial dose (0.125 mg) at the study site on the day of randomization. Dosing of study drug continued at 0.125 mg 3 times daily (TID; every 6 to 8 hours) with food. Dose increases could occur in 0.125-mg increments every 72 hours at the discretion of the Investigator up to a maximum allowable dose of 6 mg TID. Subjects received oral treprostinil as 0.125, 0.25, 1.0, or 2.5 mg sustained-release osmotic tablets (maximum dose 6 mg TID) or matching placebo. Doses of study drug were to be increased in the absence of dose-limiting drug-related adverse events (AEs) to ensure that each subject received the optimal dose throughout the study. Subjects returned for visits at Weeks 6, 12, 18, and 24. Subjects who terminated study drug early were asked to complete all remaining study visits. The study had an adaptive design where the maximum allowable dose was 2 mg until the Data Monitoring Committee had confirmed a satisfactory safety profile. After this confirmation, the maximum allowable dose was increased to 4 mg TID. This occurred after 45 subjects had been enrolled. A subsequent Data Monitoring Committee meeting, which occurred after 75 subjects had been enrolled, increased the maximum allowable dose to 6 mg TID.

Efficacy assessments consisted of 6-Minute Walk Distance (6MWD), blood collection for N-terminal pro-brain natriuretic peptide (NT-proBNP) levels, clinical worsening, WHO Functional Class (FC), Borg dyspnea score, glycated hemoglobin (HbA1c), and Kansas City Cardiomyopathy Questionnaire (KCCQ).

Safety assessments consisted of AEs, physical examinations, vital signs, 12-lead electrocardiograms (ECGs), echocardiograms (ECHOs), heart failure signs and symptoms, pregnancy testing, clinical laboratory tests, hospitalizations due to cardiopulmonary indication, and worsening heart failure as demonstrated by outpatient administration of intravenous (IV) diuretics. Subjects could have optionally provided samples for the evaluation of biomarkers and pharmacogenomics.

Subjects that completed the 24-week treatment period on study drug were permitted to enter the open-label extension study (Study TDE-HF-302).

The study was discontinued by the Sponsor on 14 October 2019 due to slow enrollment. As only a small portion of the anticipated total subjects had been enrolled, with many terminating early due to the study termination, there was a limited ability to explore the effect of oral treprostinil in this indication in this study.

ELIGIBILITY:
Inclusion Criteria:

1. The subject voluntarily gave informed consent to participate in the study.
2. The subject was 18 to 85 years of age (inclusive) at Screening (ie, date of providing written informed consent).
3. A subject could qualify if they had undergone a right heart catheterization (RHC) within 180 days of Baseline.
4. The subject had a diagnosis of heart failure with a left ventricular ejection fraction (LVEF) ≥45% by ECHO completed during Screening (prior to randomization).
5. The subject's baseline 6MWD was at least 150 meters.
6. The subject had pulmonary function tests conducted within 6 months of Screening or during the Screening Phase.
7. Subjects on a chronic medication for heart failure were on a stable dose for ≥30 days prior to randomization.
8. In the opinion of the Investigator, the subject was able to communicate effectively with study personnel, and was considered reliable, willing, and likely to be cooperative with protocol requirements, including attending all study visits.
9. Women of childbearing potential, including any female who had experienced menarche and who had not undergone successful surgical sterilization or was not postmenopausal, must have practiced true abstinence from intercourse when it was in line with their preferred and usual lifestyle, or have used 2 different forms of highly effective contraception for the duration of the study, and for at least 30 days after discontinuing study drug. Male subjects with a partner of childbearing potential must have used a condom during the length of the study, and for at least 48 hours after discontinuing study drug.
10. Subjects on chronic medications (eg, inhaled corticosteroids, long-acting beta2 adrenergic agonist, long acting muscarinic antagonists, combination inhaled drugs, anti-inflammatory drugs, oral/parenteral corticosteroids, or biologic agents) for any underlying respiratory condition were on a stable dose for ≥30 days prior to randomization.

Exclusion Criteria:

1. The subject was pregnant or lactating.
2. In the opinion of the Principal Investigator, the subject had a primary diagnosis of PH other than WHO Group 2 PH.
3. The subject had shown intolerance or significant lack of efficacy to a prostacyclin or prostacyclin analogue that resulted in discontinuation of therapy or inability to effectively titrate that therapy.
4. The subject had received any approved pulmonary arterial hypertension (PAH) therapies within 30 days of randomization. Chronic use of an approved phosphodiesterase type 5 inhibitor (PDE5-I) was allowed as long as the subject has been on a stable dose for at least 90 days prior to randomization and had a RHC confirming the parameters necessary for inclusion in the study after being on a stable PDE5-I dose for at least 30 days.
5. The subject had been hospitalized for a cardiopulmonary indication within 30 days of randomization.
6. The subject had a myocardial infarction within 90 days of randomization.
7. The subject had cardiac resynchronization therapy within 90 days of randomization or anticipated resynchronization therapy during the study treatment period.
8. The subject had liver function tests greater than 3 times the upper limit of normal at Screening, clinically significant liver disease/dysfunction, known Child-Pugh Class C hepatic disease, or noncirrhotic portal hypertension.
9. The subject had uncontrolled systemic hypertension, systolic blood pressure <100 mmHg, or a resting heart rate >100 beats per minute at Baseline.
10. The subject had known genetic hypertrophic cardiomyopathy, sarcoidosis, or cardiac amyloidosis.
11. The subject had a known history of any LVEF less than 40% by ECHO within 3 years of randomization. Note: a transient decline in LVEF below 40% that occurred and recovered more than 6 months before the start of Screening and was associated with an acute intercurrent condition (eg, atrial fibrillation) was allowed.
12. The subject had hemodynamically significant valvular heart disease as determined by the Investigator, including: greater than mild aortic and/or mitral stenosis or severe mitral and/or aortic regurgitation (>Grade 3)
13. The subject had a Body Mass Index >45 kg/m^2.
14. The subject had any musculoskeletal disorder, or had any other condition that limited ambulation.
15. The subject had end-stage renal disease requiring/receiving dialysis.
16. The subject participated in an investigational drug or device study within 30 days prior to the first dose of study drug.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-12-03 (Actual); Study Completion 2019-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mardi Gomberg-Maitland, MD, Principal Investigator — George Washington University
Locations (82):
- United States (82):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Banner University Medical Center Phoenix, Phoenix, Arizona
  - University of Arizona, Tucson, Arizona
  - VA Healthcare System of Greater Los Angeles, Los Angeles, California
  - University of California Los Angeles Pulmonary Division, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - University of California - Davis Medical Center, Sacramento, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Aurora Denver Cardiology Associates, Aurora, Colorado
  - University of Colorado Denver, Aurora, Colorado
  - National Jewish Health, Denver, Colorado
  - South Denver Cardiology, Littleton, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Medical Faculty Associates, George Washington University, Washington D.C., District of Columbia
  - Bay Area Cardiology Associates, Brandon, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - St. Vincent's Lung, Sleep, and Critical Care Specialists, Jacksonville, Florida
  - Central Florida Pulmonary Group, P.A., Orlando, Florida
  - Florida Hospital, Orlando, Florida
  - University of South Florida; Tampa General Hospital, Tampa, Florida
  - Cleveland Clinic of Florida, Weston, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Augusta University, Augusta, Georgia
  - Piedmont Physicians Georgia Lung, Austell, Georgia
  - WellStar Medical Group, Marietta, Georgia
  - University of Illinois at Chicago Hospital, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - OSF HealthCare, Peoria, Illinois
  - Indiana University Health Methodist Research Institute, INC, Indianapolis, Indiana
  - Community Physician Network, Heart and Vascular Care, Indianapolis, Indiana
  - Saint Vincent Hospital and Health Services, Indianapolis, Indiana
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Iowa Heart Center, West Des Moines, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - University of Louisville Physicians Outpatient Center, Louisville, Kentucky
  - Chest Medicine Associates, South Portland, Maine
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Brighton, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Spectrum Health Medical Group, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - St. Luke's Hospital, Chesterfield, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Barnabas Health Lung Center, Newark, New Jersey
  - Albany Medical College, Albany, New York
  - Mount Sinai Medical Center, New York, New York
  - Pulmonary Health Physicians, PC, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Asheville Cardiology Associates, Asheville, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Pinehurst Medical Clinic, Pinehurst, North Carolina
  - The Lindner Research Center The Christ Hospital Health Network, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - The Oregon Clinic, Portland, Oregon
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - AnMed Health Pulmonary and Sleep Medicine, Anderson, South Carolina
  - VitaLink Research - Anderson, Anderson, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Stern Cardiovascular Foundation, Germantown, Tennessee
  - Summit Medical Group, Knoxville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Houston Methodist Research Institute, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Intermountain Medical Center, Murray, Utah
  - Inova Heart and Vascular Institute, Falls Church, Virginia
  - Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
  - Carilion Clinic, Roanoke, Virginia
  - Providence Medical Research Center, Spokane, Washington
  - West Virginia University Hospital, Morgantown, West Virginia
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Treprostinil | Placebo
Started | 41 | 43
Completed | 25 | 27
Not Completed | 16 | 16
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Study Terminated by Sponsor | 12 | 15
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Treprostinil | Placebo | Total
Number analyzed (Participants) | 41 | 43 | 84
Age, Continuous [Median (Full Range); unit: years] | 74.0 [53 to 85] | 74.0 [46 to 82] | 74.0 [46 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 31 | 58
  Male | 14 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 39 | 43 | 82
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 7 | 8
  White | 40 | 36 | 76
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Etiology of HFpEF [Count of Participants; unit: Participants]
  Hypertension | 21 | 28 | 49
  Coronary artery disease | 8 | 3 | 11
  Obesity | 0 | 1 | 1
  Diabetes | 2 | 0 | 2
  Other | 10 | 11 | 21

OUTCOME MEASURES:

1. Primary Outcome: Change in 6MWD From Baseline to Week 24
Description: The intent of the 6-Minute Walk Test (6MWT) is to evaluate exercise capacity associated with carrying out activities of daily living.
Time Frame: Baseline to Week 24
Population: Safety Population
Measure: Median (Full Range); unit: meters
Arm/Group | Oral Treprostinil | Placebo
Number analyzed (Participants) | 29 | 28
meters | 21.0 [-195 to 62] | 23.3 [-140 to 104]

2. Secondary Outcome: Change in NT-proBNP Levels From Baseline to Week 24
Description: The NT-proBNP concentration is a biomarker associated with changes in right heart morphology and function.
Time Frame: Baseline to Week 24
Population: Safety Population
Measure: Median (Full Range); unit: pmol/L
Arm/Group | Oral Treprostinil | Placebo
Number analyzed (Participants) | 28 | 30
pmol/L | 9.5 [-133 to 499] | 11.5 [-231 to 172]

3. Secondary Outcome: Number of Subjects With First Clinical Worsening Event From Baseline to Week 24
Description: Clinical worsening was defined as the occurrence of any 1 of the following clinical worsening events: hospitalization due to a cardiopulmonary indication (a non-elective hospitalization lasting at least 24 hours in duration caused by clinical conditions directly related to PH and/or heart failure), outpatient administration of IV diuretics, death (all causes), decrease in 6MWD >15% from Baseline (or the subject was too ill to walk, and the cause was directly related to the disease under study) at 2 consecutive visits on different days (except Week 24).
Time Frame: Baseline to Week 24
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Treprostinil | Placebo
Number analyzed (Participants) | 41 | 43
Participants
  First Clinical Worsening Event | 6 | 5
  No clinical worsening event | 35 | 38

4. Secondary Outcome: Change in WHO FC From Baseline to Week 24
Description: The WHO functional classification ranges from I (subject's disease does not affect daily activities) to IV (subject's disease causes severe impairment).
Time Frame: Baseline to Week 24
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Treprostinil | Placebo
Number analyzed (Participants) | 41 | 43
Participants
  Baseline: WHO FC I | 1 | 1
  Baseline: WHO FC II | 19 | 17
  Baseline: WHO FC III | 21 | 24
  Baseline: WHO FC IV | 0 | 1
  Baseline: Not analyzed | 0 | 0
  Week 24: WHO FC I | 4 | 1
  Week 24: WHO FC II | 10 | 16
  Week 24: WHO FC III | 15 | 11
  Week 24: WHO FC IV | 0 | 0
  Week 24: Not analyzed | 12 | 15

ADVERSE EVENTS:
Time Frame: The Treatment Phase was 24 weeks for each subject. The study was discontinued by the Sponsor on 14 October 2019 due to slow enrollment.
Arm/Group | Oral Treprostinil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 1/43
Serious Adverse Events (participants affected / at risk) | 11/41 | 8/43
Other Adverse Events (participants affected / at risk) | 37/41 | 38/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Treprostinil (N=41) | Placebo (N=43)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 2 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Treprostinil (N=41) | Placebo (N=43)
Diarrhoea (Gastrointestinal disorders) | 19 (23) | 16 (19)
Headache (Nervous system disorders) | 22 (27) | 12 (14)
Nausea (Gastrointestinal disorders) | 13 (14) | 6 (7)
Fatigue (General disorders) | 8 (10) | 10 (13)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 9 (10)
Dizziness (Nervous system disorders) | 5 (7) | 9 (10)
Oedema peripheral (General disorders) | 5 (5) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 (10) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 7 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (8) | 4 (5)
Chest pain (General disorders) | 4 (4) | 3 (3)
Flushing (Vascular disorders) | 5 (5) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (3) | 5 (5)
Vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5)
Flatulence (Gastrointestinal disorders) | 3 (3) | 3 (3)
Hypotension (Vascular disorders) | 5 (6) | 1 (1)
N-terminal prohormone brain natriuretic peptide increased (Investigations) | 2 (2) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 1 (1)
Bronchitis (Infections and infestations) | 4 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Pain (General disorders) | 4 (4) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3)
Decreased appetite (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Weight increased (Investigations) | 4 (4) | 0 (0)
Blood creatinine increased (Investigations) | 3 (3) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Presyncope (Nervous system disorders) | 0 (0) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 3 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institution and/or Principal Investigator agree not to publish or publicly present any interim results of the study without the prior written consent of Sponsor, not to be unreasonably withheld or delayed. Institution and/or Principal Investigator further agree to provide Sponsor with drafts of any such publication or presentation for review and approval no less than 30 days prior to submission for publication or the date of public presentation.

DOCUMENTS (2):
  • Study Protocol (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/80/NCT03037580/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/80/NCT03037580/SAP_001.pdf